CLINICAL TRIAL: NCT03704584
Title: Corticosteroid(CS) Injections for the Treatment of Common Upper Extremity Pathologies, With or Without Lidocaine
Brief Title: Corticosteroid(CS) + Lido or Corticosteroid(CS) Alone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment and study activities were initially suspended due to COVID-19. The investigator has also left Emory and the study will not resume.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Charles A Daly, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104900
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Tenosynovitis
Keywords: orthopedic disorders; corticosteroids(CS); Lidocaine; Injections
MeSH Terms: conditions — Tenosynovitis; Musculoskeletal Diseases | interventions — Methylprednisolone Acetate; Triamcinolone Acetonide; Control Groups; Adrenal Cortex Hormones; Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized, unblinded controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (corticosteroid injection plus lidocaine) (Active Comparator): Treatment Group (corticosteroid injection plus lidocaine) subjects will receive (Methylprednisolone acetate injectable suspension and Lidocaine HCl) for their upper extremity condition
  Interventions: Drug: Treatment Group: Corticosteroid injection; Drug: Treatment Group: Lidocaine
- Control Group (corticosteroid alone) (Other): Control Group (corticosteroid alone) subjects will receive (Methylprednisolone acetate injectable suspension) for their upper extremity condition
  Interventions: Drug: Control Group (corticosteroid alone)

INTERVENTIONS:
Drug: Treatment Group: Corticosteroid injection — Subjects will receive a corticosteroid injection that is 40 mg/mL injection of Methylprednisolone or 40mg/mL injection of methylacetate injectable suspension or 40 mg/mL triamcinolone.
  Other Names: depo-medrol; kenalog
  Arms: Treatment Group (corticosteroid injection plus lidocaine)
Drug: Control Group (corticosteroid alone) — Control Group (corticosteroid alone) subjects will receive (40 mg/mL injection of Methylprednisolone acetate injectable suspension or 40 mg/mL triamcinolone) .
  Other Names: Methylprednisolone acetate injectable suspension
  Arms: Control Group (corticosteroid alone)
Drug: Treatment Group: Lidocaine — Subjects will receive an injection of lidocaine (1% lidocaine HCl).
  Other Names: Xylocaine
  Arms: Treatment Group (corticosteroid injection plus lidocaine)

SUMMARY:
The clinical trial is a randomized control trial to compare the efficacy of a combined lidocaine and corticosteroid (CS) injection versus a corticosteroid injection (CS) alone on pain, range of motion, and patient reported outcomes for the treatment of common upper extremity tendinopathies and nerve entrapments that are often treated with a combination of these injectates.

DETAILED DESCRIPTION:
A tendon is a type of tissue that connects your muscles to your bones. These tissues help control actions such as running, jumping, grasping, and lifting. Without tendons it would be difficult to control the movement of your body. A protective layer known as synovium covers tendons. This sheath produces fluid, which keeps the tendon lubricated and moving properly. Inflammation or swelling of the sheath is known as tendon sheath inflammation or tenosynovitis. This condition is often treated with an injection into or around the sheath. This injection often consists of a corticosteroid with or without lidocaine. Corticosteroid(CS) are drugs that decrease inflammation and are given for a number of orthopaedic conditions to decrease symptoms of the underlying disease. Lidocaine is also a drug that blocks the pain response, although it only blocks it momentarily. The study aims to determine if corticosteroid injection alone is as effective as corticosteroid combined with lidocaine for the relief of tenosynovitis of the upper extremity.

The study plans to enroll 1000 pts with tendinopathies of upper extremities and nerve entrapments and will be followed up in clinic 2 weeks and 6 weeks after the injection. During the clinic visits the Visual Analog Scale for pain (VAS-pain), range of motion (ROM), strength, and patient reported outcome data will be collected and any complications will be noted. Patients will also utilize a pain journal to track VAS-pain over the first 7 post-injection days.

ELIGIBILITY:
Inclusion Criteria:

* All adult clinical patients of Emory upper extremity surgeons undergoing injection for treatment of the following who are willing to participate in the study will be included in the study: Tenosynovitis of the upper extremity, including but not limited to, the shoulder, biceps, elbow, wrist, thumb, carpometacarpal, midcarpal, elbow, and small joints of the hand.
* Between the ages of 18 years and 95 years.
* For trigger finger: patients with a diagnosis of stenosing tenosynovitis based on a history of triggering and the presence of tenderness over the A1 pulley upon clinical examination. All patients, based on the Quinnell grading of trigger finger will be included.

Exclusion Criteria:

* Patients who are minors, vulnerable subjects, or who are not willing to consent to participate in the study.
* Allergies to glucocorticoids, current daily use of glucocorticoids or strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, and meperidine), severe diabetic neuropathy of the hand influencing pain perception, rheumatoid arthritis, and neurological or psychiatric diseases, potentially influencing pain perception.
* Subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Daly, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic A, Clifton Road Clinic, Atlanta, Georgia
  - 12 Executive Park Drive, Atlanta, Georgia
  - Emory Healthcare Orthopaedics and Spine Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between May 2019 and January 2020.
Pre-assignment Details: 62 individuals were consented to participate in the study and 61 individuals of these took part in the study with a total of 74 digits randomized and injected in this study. Patients were assigned to treatment groups by means of randomizing the affected unit(s) they contributed to the study.
Units Other Than Participants: digits
Groups:
- Treatment Group (Corticosteroid Injection Plus Lidocaine): Treatment Group (corticosteroid injection plus lidocaine) subjects will receive (Methylprednisolone acetate injectable suspension and Lidocaine HCl) for their upper extremity condition for their upper extremity condition
  Treatment Group (corticosteroid injection plus lidocaine): Subjects will receive (corticosteroid injection plus lidocaine) that is (40 mg/mL injection of Methylprednisolone or 40mg/mL injection of methylacetate injectable suspension or 40 mg/mL triamcinolone and 1% lidocaine HCl).
Period: Overall Study
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Started | 36; 43 digits | 26; 31 digits
Completed | 35; 42 digits | 26; 31 digits
Not Completed | 1; 1 digits | 0; 0 digits
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 62 individuals were consented to participate, and 74 digits were randomized and injected as a part of this study. One individual with one digit withdrew from the study after injection. 61 individuals completed the study, and 73 digits are available for analysis.
Units Other Than Participants: Digits
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone) | Total
Number analyzed (Participants) | 35 | 26 | 61
Number analyzed (Digits) | 42 | 31 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.00 (13) | 68 (11) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 19 | 12 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 24 | 20 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 26 | 61
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29 (5) | 32 (9) | 30.6 (7.1)
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 0 | 1 | 1
  Quit > 3 months prior | 8 | 5 | 13
  Never a smoker | 27 | 20 | 47
Comorbidities [Count of Participants; unit: Participants]
  Psychological Diagnoses (Anxiety, Depression, PTSD, Bipolar Disorder) | 5 | 5 | 10
  Diabetes | 6 | 5 | 11
  Osteoarthritis | 7 | 5 | 12
  Inflammatory Arthritis | 0 | 1 | 1
Quinnell grading system [Count of Participants; unit: Participants] — The Quinnell grading system is used to assess clinical severity of trigger finger (TF). According to this classification, TF fingers are rated as follows: 0, normal movement of the digit; 1, uneven movement; 2, actively correctable locking of the digit; 3, passively correctible locking; and 4, fixed deformity.
  Participants
    0 | 2 | 2 | 4
    1 | 11 | 9 | 20
    2 | 13 | 9 | 22
    3 | 2 | 1 | 3
    4 | 1 | 1 | 2
    Not recorded | 6 | 4 | 10
History of Prior Finger Injections [Count of Participants; unit: Participants]
  Right | 22 | 21 | 43
  Left | 13 | 5 | 18
Finger Injected [Count of Participants; unit: Participants]
  Thumb | 10 | 5 | 15
  Index | 7 | 2 | 9
  Middle | 9 | 13 | 22
  Ring | 5 | 4 | 9
  Little | 4 | 2 | 6
Dominant Hand Injected [Count of Participants; unit: Participants] | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: 10 Point Likert Scale of Pain Scores Before the Injection and After the Injection and During Follow up in the Corticosteroid Plus Lidocaine Group as Compared to the Corticosteroid Alone Group
Description: Pain will be assessed with a 10-point scale (0: no pain, 10: highest amount of pain) of anticipated pain and anxiety before injection and a 10-point pain scale of the pain of the needle, medication, overall pain and anxiety after the injection was administered to the participants.
Time Frame: Pre injection, Post injection day, 2 weeks and at 6 weeks
Population: There was a total of 62 participants enrolled in the study. One patient withdrew after injection and has been excluded from analysis. Only 61 participants contributed data to the summary assessment. 35 in the treatment group and 26 in the control group. The total number of units (digits) analyzed was 73 (digits). 42 digits were analyzed in the treatment group and 31 digits in the control group.
  Due to time constraints at follow up study visits, data was not collected for 2 and 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Digits
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 35 | 26
Number analyzed (Digits) | 42 | 31
score on a scale
  Pre-Injection: How painful do you think the injection will be? | 5.9 (2.3) | 5.4 (2.6)
  Pre-Injection: How painful do you think it will be 1-minute after the injection? | 4.4 (2.6) | 3.2 (2.7)
  Pre-Injection: How nervous are you about the injection? | 4.0 (3.5) | 3.5 (3.3)
  Post-Injection: Actual pain of the needle | 4.3 (3.1) | 4.2 (2.9)
  Post-Injection: Actual pain of the medication | 4.7 (3.2) | 4.3 (2.8)
  Post-Injection: Actual pain 1-minute after the injection | 1.7 (2.2) | 1.7 (2.2)
  2 weeks post intervention: number analyzed (Participants) | 0 | 0
  2 weeks post intervention: number analyzed (Digits) | 0 | 0
  6 weeks post intervention: number analyzed (Participants) | 0 | 0
  6 weeks post intervention: number analyzed (Digits) | 0 | 0

2. Primary Outcome: Visual Analog Pain Scale (VAS-pain) Daily Until Post-injection Day 7
Description: Participants were instructed to log their pain twice daily (morning and night) using a VAS pain scale of 0-10 (0: no pain, 10: highest amount of pain) for the first 7 days after injection. Participants were instructed to bring that pain journal to their 2-week visit. Average daily scores are presented.
Time Frame: Post injection day (1-7), 2 weeks and at 6 weeks post intervention
Population: 32 participants were seen for a 2-week follow-up and pain journal were collected. Other patients were non compliant with completion of their pain journal or were not seen at 2-weeks. Due to time constraints at follow up study visits, no other data was collected at 2 and 6 weeks post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 20 | 12
score on a scale
  Post injection day 1 | 3.7 (2.2) | 3.7 (3.0)
  Post injection day 2 | 2.2 (2.0) | 3.0 (2.9)
  Post injection day 3 | 1.7 (1.9) | 2.6 (2.6)
  Post injection day 4 | 1.1 (1.5) | 2.2 (2.0)
  Post injection day 5 | 1.0 (1.4) | 2.0 (2.2)
  Post injection day 6 | 0.69 (1.1) | 1.5 (1.8)
  Post injection day 7 | 0.58 (0.95) | 1.6 (1.9)
  2 weeks post intervention: number analyzed (Participants) | 0 | 0
  6 weeks post intervention: number analyzed (Participants) | 0 | 0

3. Primary Outcome: Quick Disabilities of Arm, Shoulder and Hand (QuickDASH) Scores at Follow up in the Corticosteroid Plus Lidocaine Group as Compared to the Corticosteroid Alone Group
Description: The domains explored by the Quick DASH are: (1) physical arm, shoulder or hand activity problems (6 items); (2) severity of pain and tingling (2 items); (3) social activities, work, and sleep (3 items). Each item has five response options, ranging from 1, ''no difficulty or no symptom,'' to 5, ''unable to perform activity or very severe symptom.'' If at least 10 of the 11 items are completed, a score ranging from 0 (no disability) to 100 (most severe disability) can be calculated [(sum of n responses/n) - 1] x 25.the effect size and the percentage of patients reaching Minimal Clinical Important Improvement was determined.
Time Frame: 2 weeks and at 6 weeks post intervention
Population: Due to time constraints at study visits, the decision was made to not administer the QuickDASH surveys
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Patient-Rated Wrist Evaluation (PRWE) Score at Follow up in the Corticosteroid Plus Lidocaine Group as Compared to the Corticosteroid Alone Group
Description: The Patient-Related Wrist Evaluation is a score for the measurement of pain and function after injury to the wrist. The PRWE is a 15-item questionnaire that allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of 2 subscales Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0 Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0. Total Score = Sum of pain+ function scores (Best Score = 0, Worst Score = 100).
Time Frame: 2 weeks and at 6 weeks post intervention
Population: Due to time constraints at study visits, the decision was made to not administer the PRWE questionnaire.
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: American Shoulder and Elbow Surgeons Shoulder Score (ASES) at Follow up in the Corticosteroid Plus Lidocaine Group as Compared to the Corticosteroid Alone Group
Description: The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is a mixed outcome reporting measure, applicable for use in all patients with shoulder pathology for the assessment of shoulder function. The ASES questionnaire is composed of 17 questions. The questions focus on joint pain, instability, and activities of daily living. It is a 100 point scale (Pain scale= 50 points, 10 activities of daily living = 50 points).Score range: Pain subscale 0-50 ASES points; function/disability subscale 0-50 ASES points. Total score 0-100 ASES points (0 = worse pain and functional loss/disability)
Time Frame: 2 weeks and at 6 weeks post intervention
Population: Due to time constraints at study visits, the decision was made to not administer the ASES questionnaire.
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Short Form Health Survey (SF-12) Scores at Follow up in the Corticosteroid Plus Lidocaine Group as Compared to the Corticosteroid Alone Group
Description: The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. SF-12 is a standardized self-report questionnaire that assesses mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for each component ranging from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Time Frame: 2 weeks and at 6 weeks post intervention
Population: Due to time constraints at study visits, the decision was made to not administer the SF-12 survey.
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Patients With Subsequent Reinjection and Surgical Operation
Description: The number of patients with subsequent reinjection and surgical operation was collected during follow up.
Time Frame: End of follow up (6 weeks post intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
Number analyzed (Participants) | 35 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Data collected during 6 weeks follow up post intervention (post injection).
Arm/Group | Treatment Group (Corticosteroid Injection Plus Lidocaine) | Control Group (Corticosteroid Alone)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/26
Other Adverse Events (participants affected / at risk) | 0/35 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT03704584/Prot_SAP_000.pdf